CLINICAL TRIAL: NCT04844359
Title: Development and Validation of a Prognostic Transcriptomic Signature for Chronic Hypersensitivity Pneumonitis
Brief Title: A Prognostic Transcriptomic Signature for Chronic Hypersensitivity Pneumonitis
Acronym: PREDICT-HP
Status: Active, not recruiting | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: University of California, Davis (Other); Mayo Clinic (Other); University of Chicago (Other); University of Texas Southwestern Medical Center (Other); University of Arizona (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Evans Fernandez Perez, Associate Professor, National Jewish Health
Other Study IDs: R01HL148437 (NIH)
Record Dates: First submitted 2021-03-30; First posted 2021-04-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hypersensitivity Pneumonitis
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Up to 150 patients with hypersensitivity pneumonitis will be enrolled at 7 clinical centers across the United States. Patients will be followed for 24 months to determine if biomarkers in the blood can predict disease progression.

DETAILED DESCRIPTION:
Hypersensitivity pneumonitis is an immunologically mediated form of lung disease, resulting from inhalation exposure to a large variety of antigens. For unknown reasons, a subgroup of patients with HP without a known inciting antigen exposure develops chronic disease with progressive pulmonary fibrosis (the leading cause of death). Accurately identifying patients at risk of disease progression is necessary for prognosis and therapy.

Enrolled subjects will be followed for 24 months and complete 5 visits to one of the study centers. Blood biomarkers will be collected in addition to other clinical data to determine if these biomarkers can predict disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hypersensitivity pneumonitis
* Age 18 through 85 years.
* Diagnosis of chronic hypersensitivity pneumonitis by HRCT
* Able to understand and sign a written informed consent form.
* Able to understand the importance of adherence to the study protocol and willing to follow all study requirements

Exclusion Criteria:

* Not a suitable candidate for enrollment or unlikely to comply with the requirements of this study
* Known explanation for the interstitial lung disease
* Clinical diagnosis of any connective tissue disease
* Listed or expected to receive a lung transplant within 4 months from enrollment
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of men and women aged 18 to 85 years old with a diagnosis of chronic hypersensitivity pneumonitis.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to absolute FVC (percent predicted) decline ≥10 percent | Up to 24 months
Time to absolute DLCO (percent predicted) decline ≥10 percent | Up to 24 months
Time to relative FVC (percent predicted) decline ≥10 percent | Up to 24 months
Time to relative DLCO (percent predicted) decline ≥10 percent | Up to 24 months
Time to relative DLCO (percent predicted) decline ≥15 percent | Up to 24 months
Time to first adjudicated acute chronic hypersensitivity pneumonitis exacerbation | Up to 24 months
Need for a new course of oral or intravenous steroids | Up to 24 months
Time to death from any cause | Up to 24 months
Change from baseline in St. George's Respiratory Questionnaire total score at month 6 | 6 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in St. George's Respiratory Questionnaire total score at month 12 | 12 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in St. George's Respiratory Questionnaire total score at month 18 | 18 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in St. George's Respiratory Questionnaire total score at month 24 | 24 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using University of California San Diego Shortness of Breath Questionnaire at month 6 | 6 months
  Scores range from 0 to 120, with higher scores indicating greater breathlessness.
Change from baseline in dyspnea using University of California San Diego Shortness of Breath Questionnaire at month 12 | 12 months
  Scores range from 0 to 120, with higher scores indicating greater breathlessness.
Change from baseline in dyspnea using University of California San Diego Shortness of Breath Questionnaire at month 18 | 18 months
  Scores range from 0 to 120, with higher scores indicating greater breathlessness.
Change from baseline in dyspnea using University of California San Diego Shortness of Breath Questionnaire at month 24 | 24 months
  Scores range from 0 to 120, with higher scores indicating greater breathlessness.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire symptoms score at month 6 | 6 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire symptoms score at month 12 | 12 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire symptoms score at month 18 | 18 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire symptoms score at month 24 | 24 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire activity score at month 6 | 6 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire activity score at month 12 | 12 months
Change from baseline in dyspnea using St. George's Respiratory Questionnaire activity score at month 18 | 18 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire activity score at month 24 | 24 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire impact score at month 6 | 6 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire impact score at month 12 | 12 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire impact score at month 18 | 18 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in dyspnea using St. George's Respiratory Questionnaire impact score at month 24 | 24 months
  The total score ranges from 0 to 100, with higher scores indicating worse health-related quality of life.
Change from baseline in CT visual (≥10 percent) score at month 12 | 12 months
  Visual scores range from 0 to 100, with higher scores indicating more lung fibrosis.
Change from baseline in CT visual (≥10 percent) score at month 24 | 24 months
  Visual scores range from 0 to 100, with higher scores indicating more lung fibrosis.
Change from baseline in CT quantitative (≥3.4) score at month 12 | 12 months
  CT quantitative scores range from 0 to no upper limits, with higher scores indicating more lung fibrosis.
Change from baseline in CT quantitative (≥3.4) score at month 24 | 24 months
  CT quantitative scores range from 0 to no upper limits, with higher scores indicating more lung fibrosis.
Change from baseline in 6-min walk distance at month 6 | 6 months
Change from baseline in 6-min walk distance at month 12 | 12 months
Change from baseline in 6-min walk distance at month 18 | 18 months
Change from baseline in 6-min walk distance at month 24 | 24 months
Rate of decline in FVC (percent predicted) over 24 months | Up to 24 months
Rate of decline in FVC (ml) over 24 months | Up to 24 months
Rate of decline in DLCO (percent predicted) over 24 months | Up to 24 months
Rate of decline in DLCO (mmol/min/kpa) over 24 months | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Evans Fernández, MD, MS, Principal Investigator — National Jewish Health
Locations (7):
- United States (7):
  - University of Arizona, Tucson, Arizona
  - University of California Davis, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah